CLINICAL TRIAL: NCT05882929
Title: The Effect of Distraction Methods on Pain Level and Physiological Parameters in the Postoperative Period of Pediatric Patients Undergoing Outpatient Surgery: A Randomized Controlled Study
Brief Title: The Effect of Distraction in the Postoperative Period of Pediatric Patients Undergoing Outpatient Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sevinc Akkoyun, assistant professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021/45
Record Dates: First submitted 2022-12-03; First posted 2023-05-31 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative; Surgery; Child, Only
Keywords: Pain; Surgery; Pediatric; Postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled trial. In this parallel group study, there will be two intervention groups (watching cartoons and ball squeezing) and a control group.
Who Masked: Participant
Masking Description: Single (participant, outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experiment 1: Watching Cartoons (Experimental): Watching Cartoon Movies will be performed after the child comes to the service after the operation and prepares for the postoperative period (taking vital signs, putting on clothes, controlling bleeding, telling the feeding time, etc.). Interventions will be implemented for a total of 15 minutes. Physiological Parameters Follow-up Form and Wong-Baker Faces Pain Scale will be filled in before the interventions are applied, 10 minutes during the intervention and 5 minutes after the intervention is completed.
  Interventions: Other: Watching Cartoons
- Experiment 1: ball spin (Experimental): ball squeezing will be applied after the child comes to the service after the operation and the postoperative period preparation is made (taking the vital signs, putting on the clothes, controlling the bleeding, telling the feeding time, etc.). Interventions will be implemented for a total of 15 minutes. Physiological Parameters Follow-up Form and Wong-Baker Faces Pain Scale will be filled in before the interventions are applied, 10 minutes during the intervention and 5 minutes after the intervention is completed.
  Interventions: Other: ball spin
- Control (No Intervention): In the control group, the 10th and 20th minute physiological parameters and Wong-Baker Faces Pain Scale will be evaluated after the child comes to the service after the operation and is prepared for the postoperative period (taking vital signs, putting on clothes, controlling bleeding, telling the feeding time, etc.).

INTERVENTIONS:
Other: Watching Cartoons — The cartoon will be watched after the child comes to the service after the operation and the postoperative period is prepared (taking the vital signs, putting on the clothes, controlling the bleeding, telling the feeding time, etc.).
  Arms: Experiment 1: Watching Cartoons
Other: ball spin — ball squeezing will be applied after the child comes to the service after the operation and after the postoperative period preparation is made (taking the vital signs, dressing the clothes, controlling the bleeding, telling the feeding time, etc.).
  Arms: Experiment 1: ball spin

SUMMARY:
The aim of the study is to examine the effects of distraction methods such as watching cartoons and ball squeezing on the level of pain and physiological parameters in the postoperative period in children aged 6-12 years who have outpatient surgery. The research is a randomized controlled trial. The sample number was determined as 40 children (total 120) in each group. Information Form, Physiological Parameters Follow-up Form, Wong-Baker Faces Pain Scale will be used to collect research data. In the initiative group, two attempts will be implemented, namely watching cartoons and squeezing the ball. Interventions will be implemented for a total of 15 minutes. Physiological Parameters Follow-up Form and Wong-Baker Faces Pain Scale will be filled in before the interventions are applied, 10 minutes during the intervention and 5 minutes after the intervention is completed. In the control group, the 10th and 20th minute physiological parameters and the Wong-Baker Faces Pain Scale will be evaluated after the child comes to the service after the operation and is prepared for the postoperative period (taking vital signs, putting on clothes, controlling bleeding, telling the feeding time, etc.). In the analysis of study data; chi-square test for descriptive statistics, chi-square test for repeated measurements, single factor analysis of variance, Mann-Whitney U test and Friedman will be used. In the study, values at the p<0.05 level were considered statistically significant.

DETAILED DESCRIPTION:
The aim of the study is to examine the effects of distraction methods such as watching cartoons and ball squeezing on the level of pain and physiological parameters in the postoperative period in children aged 6-12 years who have outpatient surgery. The research is a randomized controlled trial. The sample number was determined as 40 children (total 120) in each group. Information Form, Physiological Parameters Follow-up Form, Wong-Baker Faces Pain Scale will be used to collect research data. In the initiative group, two attempts will be implemented, namely watching cartoons and squeezing the ball. Interventions will be implemented for a total of 15 minutes. Physiological Parameters Follow-up Form and Wong-Baker Faces Pain Scale will be filled in before the interventions are applied, 10 minutes during the intervention and 5 minutes after the intervention is completed. In the control group, the 10th and 20th minute physiological parameters and the Wong-Baker Faces Pain Scale will be evaluated after the child comes to the service after the operation and is prepared for the postoperative period (taking vital signs, putting on clothes, controlling bleeding, telling the feeding time, etc.). In the analysis of study data; chi-square test for descriptive statistics, chi-square test for repeated measurements, single factor analysis of variance, Mann-Whitney U test and Friedman will be used. In the study, values at the p<0.05 level were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years
* Children with day surgery surgery
* Children with American Society of Anesthesiologists classification (ASA) I-II (ASA score is given in the preoperative period by the anesthesiologist)
* Parents who volunteered to participate in the study
* Turkish speaking children

Exclusion Criteria:

* Children who have had previous surgery
* Children with the American Society of Anesthesiologists classification (ASA) III
* Children with congenital anomalies, psychiatric, neurological and chronic diseases

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
pain level of children | Just before the interventions and 5 minutes after the intervention
  Wong Baker Pain Faces Scale mean score Wong-Baker Pain Faces Scale is widely used with people ages three and older, not limited to children. This self-assessment tool must be understood by the patient, so they are able to choose the face that best illustrates the physical pain they are experiencing. It is a tool to be used by a third person, parents, healthcare professionals, or caregivers, to assess the patient's pain. The scale is 0-10 scale. The six illustrated faces on the cards show a range of emotions, from a smiling face (0 'no pain) to a crying face (10 "worst pain"). 0 indicates no pain, 10 indicates the most severe pain. It is measured before, at the 10th minute and after the intervention.
physiological parametres of the child: body temperature level | Just before the interventions and 5 minutes after the intervention
  body temperature change
physiological parametres of the child: peak heart rate | Just before the interventions and 5 minutes after the intervention
  heart rate change
physiological parametres of the child: respiratory rate | Just before the interventions and 5 minutes after the intervention
  respiratory rate change
physiological parametres of the child: oxygen saturation (SpO2) | Just before the interventions and 5 minutes after the intervention
  SpO2 level change

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Tas Arslan, professor, Study Director — Selcuk University; Mehmet Sarıkaya, Doctor, Study Chair — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The effect of distraction methods on the postoperative period of pediatric patients undergoing outpatient surgery
Supporting Information: Study Protocol
Time Frame: December 2022-July 2023 (7 months)